CLINICAL TRIAL: NCT04404387
Title: A Multicentre Concealed-Allocation Parallel-Group Blinded Randomized Controlled Trial to Ascertain the Effect of High-Dose Intravenous Vitamin C Compared to Placebo on Mortality or Persistent Organ Dysfunction at 28 Days in Septic Intensive Care Unit Patients
Brief Title: Lessening Organ Dysfunction With VITamin C in Septic ARDS
Acronym: LOVIT ARDS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP200019; 2019-003350-80 (Registry Identifier: IDRCB); 2020-003923-40 (EudraCT Number)
Record Dates: First submitted 2020-05-19; First posted 2020-05-27 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Septic; Acute Respiratory Distress Syndrome
Keywords: Septic; Acute respiratory distress syndrome; Vitamin C
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): vitamin C 50 mg/kg every 6 hours for 96 hours.
  Interventions: Drug: Administration of vitamin C
- Control arm (Placebo Comparator): Placebo administration
  Interventions: Drug: Administration of placebo

INTERVENTIONS:
Drug: Administration of vitamin C — The intervention is intravenous vitamin C administered in bolus doses of 50 mg/kg mixed in a 50-mL solution of either dextrose 5% in water (D5W) or normal saline (0.9% NaCl), during 30 to 60 minutes or more for participants over 120 kg not to exceed 100 mg/minute, every 6 hours for 96 hours (i.e. 200 mg/kg/day and 16 doses in total).
  The other name of the drug: Ascorbic acid.
  Other Names: Administration of Ascorbic acid
  Arms: Experimental arm
Drug: Administration of placebo — Administration of placebo. Patients (in the control arm) will receive dextrose 5% in water (D5W) or normal saline (0.9% NaCl) in a volume to match the vitamin C. Placebo will be infused over 30 to 60 minutes or more for participants over 120 kg not to exceed 100 mg/minute as per the infusion instructions of vitamin C.
  Arms: Control arm

SUMMARY:
The primary objective of the study aims to compare the effect of high-dose intravenous vitamin C vs. placebo on a composite of death or persistent organ dysfunction - defined as continued dependency on mechanical ventilation, new renal replacement therapy, or vasopressors - assessed at 28 days on intensive care unit (ICU) patients.

As secondary objectives, the study aims:

* To compare the effect of high-dose intravenous vitamin C vs. placebo on:

  1. 6-month mortality;
  2. 6-month HRQoL;
  3. organ function (days 1, 2, 3, 4, 7, 10, 14, and 28 if in ICU);
  4. global tissue dysoxia (at baseline);
  5. oxygenation Index (FiO2 x Mean Airway Pressure/PaO2) (days 1, 2, 3, 4, 7, 10, 14, and 28 if in ICU, and if still intubated);
  6. occurrence of stage 3 acute kidney injury as defined by KDIGO (Kidney Disease: Improving Global Outcomes) criteria20;
  7. acute hemolysis as defined by:

     * clinician judgment of hemolysis, as recorded in the chart, or
     * hemoglobin drop of at least 25 g/L within 24 hours of a dose of investigational product PLUS 2 of the following:

       * reticulocyte count >2 times upper limit of normal at clinical site lab;
       * haptoglobin < lower limit of normal at clinical site lab;
       * indirect (unconjugated) bilirubin >2 times upper limit of normal at clinical site lab;
       * lactate dehydrogenase (LDH) >2 times upper limit of normal at clinical site lab.

     Severe hemolysis:

     - hemoglobin < 75 g/L AND at least 2 of the above criteria AND requires 2 units of packed red blood cells;
  8. hypoglycemia as defined as core lab-validated glucose levels of less than < 3.8 mmol/L.
* To assess baseline vitamin C levels in study participants (before the first dose of investigational product).

DETAILED DESCRIPTION:
Treatment options for sepsis complicated by ARDS are limited to antimicrobials and supportive care (intravenous fluids, vasopressors, mechanical ventilation and renal replacement therapy). Recent preliminary evidence suggests that intravenous vitamin C may be the first therapy to mitigate the dysregulated cascade of events transforming an infection into sepsis. However, definitive practice changing evidence requires a large trial powered to detect a plausible, modest, and clinically important difference in mortality.

The study LOVIT will be conducted simultaneously in Canada (country of coordination), France, the United States of America, the United Kingdom and Australia/New Zealand.The data from each country will be merged with the aim of reaching 4,000 patients globally (roughly 800 patients per country). Thus, in the context of increasing off-label use of vitamin C for sepsis and ongoing trials of vitamin C bundled with other pharmacological interventions, this study will constitute a rigorous assessment of the effect of vitamin C monotherapy on patient-important outcomes. Moreover, the French LOVIT-ARDS, part of LOVIT, will provide additional information on the specific subgroup of patients with sepsis and ARDS.

This is a prospective multicentric randomized controlled trial. Web-based randomization system available 24/7. Eligible patients will be randomized in a 1:1 ratio to vitamin C or matching placebo. The study will use permuted blocks of undisclosed and variable size and stratify randomization by site.

The study will enroll a total of at least 770 patients. Sites are expected to enroll at least 1or 2 patients per month. By enrolling 385 evaluable patients per arm, the study will have 80% power to detect a 10% absolute risk reduction (from 50% to 40%, which corresponds to a 20% relative risk reduction).

Follow-up in the study for each patient: daily during ICU stay and telephone follow-up at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years;
* Admitted to ICU with proven or suspected infection as the main diagnosis;
* Currently treated with a continuous intravenous infusion of vasopressors (norepinephrine, epinephrine, vasopressin, dopamine, phenylephrine);
* Presenting with Acute Respiratory Distress Syndrome
* Patient who has signed an informed and written consent, whenever he/she is capable of consent, if not ascent from his/her representant whenever he/she is present at time of screening for inclusion
* Affiliation to a social security system or to an universal health coverage (Couverture Maladie Universelle, CMU).
* Patients under guardianship or curatorship will be included.
* Patients in case of simple emergency (legal definition) will be included.

Exclusion Criteria:

* > 24 hours of intensive care unit (ICU) admission;
* Known Glucose-6-phosphate dehydrogenase (G6PD) deficiency;
* Pregnancy;
* Known allergy to vitamin C;
* Known kidney stones within the past 1 year;
* Received any intravenous vitamin C during this hospitalization unless incorporated in parenteral nutrition;
* Expected death or withdrawal of life-sustaining treatments within 48 hours;
* Previously enrolled in this study;
* Previously enrolled in a trial for which co-enrolment is not allowed (co-enrolment to be determined case by case).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2022-07-22 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Number of deceased participants or with persistent organ dysfunction | Both assessed at 28 days
  Defined as death or persistent organ dysfunction: continued dependency on mechanical ventilation, renal replacement therapy, or vasopressors.

SECONDARY OUTCOMES:
Vital statue at 6 months | at 6 months
  Mortality at 6 months
Quality of life assessement: EQ-5D-5L | at 6 months
  Quality of life of patients will be assessed by the questionnaire EQ-5D-5L.
  The questionnaire EQ-5D-5L essentially consists of 2 pages:
  - page1: the EQ-5D-5L descriptive system:
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box (1-digit number) next to the most appropriate statement in each of the five dimensions.
  - page 2: the EQ visual analogue scale (VAS): the EQ VAS records the patient's self-rated health on a vertical visual analogue scale.
  The 2 parts of the questionnaire can not be assessed seperately.
Daily organ function | Days 1, 2, 3, 4, 7, 10, 14, 28
  Daily organ function (SOFA score days 1, 2, 3, 4, 7, 10, 14, and 28);
Global tissue dysoxia | At baseline and days 1, 3, 7
  Global tissue dysoxia: assessed by serum lactate concentration
Occurrence of stage 3 acute kidney injury | Up to day 28
  Occurrence of stage 3 acute kidney injury as defined by KDIGO criteria
Acute hemolysis | Up to day 28
  Acute hemolysis as defined by:
  * clinician judgment of hemolysis, as recorded in the chart, OR
  * hemoglobin drop of at least 25 g/L within 24 hours of a dose of investigational product PLUS 2 of the following:
    * reticulocyte count >2 times upper limit of normal at clinical site lab;
    * haptoglobin < lower limit of normal at clinical site lab;
    * indirect (unconjugated) bilirubin >2 times upper limit of normal at clinical site lab;
    * LDH >2 times upper limit of normal at clinical site lab.
  Severe hemolysis:
  - hemoglobin < 75 g/L AND at least 2 of the above criteria AND requires 2 units of packed red blood cells.
Hypoglycemia | During the time participants receive the 16 doses of the investigational product and the 7 days following the last dose
  Hypoglycemia as defined by core lab-validated glucose levels of less than < 3.8 mmol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Djillali ANNANE, MD, PhD, Principal Investigator — Department Intensive Care Unit, Hospital Raymond Poincaré - APHP
Locations (1):
- Department Intensive Care Unit, Hospital Raymond Poincaré - APHP, Garches, France

IPD SHARING:
Plan to Share IPD: No